CLINICAL TRIAL: NCT02014142
Title: A Phase 2 Single-Masked, Randomized Study of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Brief Title: A Phase 2 Single-Masked, Randomized Study of Latanoprost PPDS in Ocular Hypertension or Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPL GLAU M1
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Group A. L-PPDS single occlusion (Experimental): Latanoprost Punctal Plug Delivery System (L-PPDS) continuous single occlusion; L-PPDS will be inserted in the lower punctum and no plug will be inserted in the upper punctum of each eye; L-PPDS will remain for a period of 14 weeks.
  Interventions: Drug: Latanoprost Punctal Plug Delivery System (L-PPDS)
- Group B. L-PPDS double occlusion (Experimental): Latanoprost Punctal Plug Delivery System (L-PPDS) continuous double occlusion; L-PPDS will be inserted in the lower punctum and non-therapeutic (NT) plug will be inserted in the upper punctum of each eye and both will remain for a period of 14 weeks.
  Interventions: Drug: Latanoprost Punctal Plug Delivery System (L-PPDS)

INTERVENTIONS:
Drug: Latanoprost Punctal Plug Delivery System (L-PPDS) — Latanoprost Punctal Plug Delivery System (L-PPDS)

SUMMARY:
Determine efficacy of the latanoprost punctal plug. Effect of configuration of L-PPDS placement on efficacy will also be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older at the time of the screening examination
2. Subject diagnosed with bilateral OAG or OH
3. Subject IOP is currently controlled (< 21 mmHg) with a topical prostaglandin or in conjunction with one other topical ocular hypotensive drug, not including any fixed-combination formulations (i.e., Cosopt, Combigan, Azarga, etc.) for at least one month or more
4. Subject who has lower and upper puncta > 0.5 mm and < 0.9 mm (pre-dilation) in both eyes
5. Subject must be able and willing to read, comprehend and give Authorization for Use/Disclosure of Health Information (HIPAA) and informed consent
6. Subject must be willing to comply with study instructions, dosing (if applicable), agree to make all office appointments, and complete the entire course of the study
7. Women of child-bearing potential must not be pregnant or lactating, must have a negative pregnancy test at screening and must be practicing an adequate method of birth control, including intrauterine device (IUD); oral, dermal ("patch"), implant or injected contraceptives; tubal ligation; or barrier methods with spermicide
8. Subject has a central corneal thickness of > 500 μm and < 600 μm in study eye
9. Subject has a BCVA or pinhole visual acuity (Snellen) of 20/100 or better in both eyes

Exclusion Criteria:

1. Subject with a history of non-response to topical prostaglandin eye drops for OAG/OH
2. Subject with angle-closure glaucoma, neovascular glaucoma, traumatic glaucoma or iridocorneal endothelium syndrome in either eye
3. Subject with a known sensitivity to latanoprost, timolol, fluorescein, topical anesthetic, silicone, any inactive ingredient of the L-PPDS or any other products required for the study procedures
4. Subject with a history of intolerance to topical beta-blocker therapy
5. Subject with > 0.8 vertical cup or completely notched optic nerve head rim in either eye
6. Subject with any functionally significant visual field loss or progressive field loss within the last year in either eye
7. Subject with a history of complications, AEs, trauma or disease in the nasolacrimal area, whether or not it was due to punctal plug wear, including but not limited to dacryocystitis, inflammation or canaliculitis in study eye
8. Subject with structural lid abnormalities (i.e., ectropion, entropion) in study eye
9. Subject with an active lid disease in either eye (i.e., moderate or severe blepharitis, meibomianitis) that requires medical treatment
10. Subject with a history of chronic/recurrent inflammatory eye disease (i.e., scleritis, uveitis, herpes keratitis) in either eye
11. Subject who would require the use of any ocular topical medication(s), an over-the counter drop(s), ointment(s) or gel(s), other than the study ocular hypotensive medication(s) in either eye during the study period
12. Subject who has had any ophthalmic surgical procedures (i.e., glaucoma laser, minimally invasive glaucoma surgery, cataract, refractive, etc.) in study eye within the last six months or will require ophthalmic surgery before completing the study
13. Subject with a history of penetrating keratoplasty in study eye
14. Subject who is incapable of instilling ocular drops into his or her eyes
15. Subject requiring the use of a contact lens in either eye at any time during the study period
16. Subject with advanced diabetic retinopathy, branch retinal vein occlusion or central retinal vein occlusion in either eye
17. Subject with a history of macular edema in either eye
18. Subject currently on any systemic medication [i.e., beta-blocker, carbonic anhydrase inhibitors, corticosteroids (including dermal), etc.], that may have an effect on the subject's IOP, or who will require its use during the study period (Note: an inhaled steroid, systemic beta-blocker or β-adrenoceptor antagonist may be permitted, providing the subject has maintained a stable dosage regimen for at least the last three months)
19. Subject contraindicated to therapy with a beta-blocker (i.e., history or presence of bradycardia, untreated congestive heart failure, untreated second- or third-degree heart block, sino-atrial block, myasthenia gravis, cardiogenic shock, history or presence of bronchial asthma, bronchial hyperreactivity, severe chronic obstructive pulmonary disease, or history of bronchospasm)
20. Subject with an uncontrolled systemic disease or a medical condition that may increase the risk associated with study participation or administration of study treatment or that may interfere with the interpretation of study results (e.g., autoimmune disease if the subject is on chronic medications and has ocular involvement; host-versus-graft disease)
21. Subject currently participating or has participated within the last 30 days prior to the start of this study in a drug, device or other investigational research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline and the primary analysis time point will be the IOP assessment at Week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Arizona Eye Center, Chandler, Arizona
  - Arizona Glaucoma Specialists, Phoenix, Arizona
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Argus Research at Cape Coral Eye Center, Cape Coral, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Indiana Universtiy - Eugene and Marilyn Glick Eye Institute Ophthalmology Center, Indianapolis, Indiana
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Chu Vision Institute, Bloomington, Minnesota
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Abrams Eye Institute, Las Vegas, Nevada
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Dr. Steven T. Simmons, Slingerlands, New York
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Phildelphia, Pennsylvania
  - University Eye Surgeons, Maryville, Tennessee
  - Total Eye Care, Memphis, Tennessee